CLINICAL TRIAL: NCT06135415
Title: A Phase 3, Multicentre, Randomised, Double-blind, Vehicle-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Tirbanibulin 10 mg/g Ointment Applied to a Treatment Field Larger Than 25 cm^2 and up to 100 cm^2 in Adult Patients With Actinic Keratosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Tirbanibulin Ointment in Adult Participants With Actinic Keratosis
Acronym: TirbAKare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-14867-33; 2023-505487-11-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Keratosis, Actinic
Keywords: Actinic Keratosis; Keratosis; Keratosis, Actinic; Precancerous condition; Neoplasms; Sun Damaged Skin; Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic; Keratosis; Precancerous Conditions; Neoplasms | interventions — tirbanibulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirbanibulin 10 mg/g (Experimental): Participants will apply tirbanibulin 10 mg/g ointment once daily for 5 consecutive days beginning on Day 1. All participants will be evaluated for efficacy, safety, and tolerability at Day 8, 15, 29, and 57. Participants who do not achieve complete clearance (CC) at Day 57 will receive a second 5-day course of the treatment. Participants receiving a second treatment course will also be evaluated for efficacy, safety, and tolerability at Day 64, 71, and 85.
  Interventions: Drug: Tirbanibulin
- Vehicle ointment (Placebo Comparator): Participants will apply vehicle ointment once daily for 5 consecutive days beginning on Day 1. All participants will be evaluated for efficacy, safety, and tolerability at Day 8, 15, 29, and 57. Participants who do not achieve CC at Day 57 will receive a second 5-day course of the treatment. Participants receiving a second treatment course will also be evaluated for efficacy, safety, and tolerability at Day 64, 71, and 85.
  Interventions: Other: Vehicle ointment

INTERVENTIONS:
Drug: Tirbanibulin — Participants will apply tirbanibulin ointment topically on the face or balding scalp with AK.
  Other Names: Klisyri®
  Arms: Tirbanibulin 10 mg/g
Other: Vehicle ointment — Participants will apply vehicle ointment topically on the face or balding scalp with AK.
  Arms: Vehicle ointment

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of tirbanibulin 10 milligrams per gram (mg/g) ointment when applied to a treatment field (TF) larger than 25 centimeter square (cm^2) and up to 100 cm^2 in adult participants with actinic keratosis (AK).

ELIGIBILITY:
Inclusion Criteria:

* Participants having a TF on the face or balding scalp (excluding lips, eyelids, and inside nostrils and ears) that contains >= 4 to less than or equal to (<=) 12 clinically typical, visible, and discrete (non-confluent) AK lesions and measures more than 25 cm2 (example, one cheek) and up to approximately 100 cm2 (example, mid face).
* Participants willing to avoid excessive sunlight or UV light exposure, including the use of tanning beds, to the face or scalp during the study.
* Women of childbearing potential (WOCBP), that is, fertile, defined as a female in the life period from menarche and until becoming post-menopausal (no menses for 12 months without an alternative medical cause) or permanently sterile (with hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least 3 months prior to screening) must have a negative urine pregnancy test using a highly sensitive method at screening and on Day 1 prior to treatment administration, be using highly effective methods of birth control for at least 30 days or 1 menstrual cycle, whichever is longer, and until at least 30 days or 1 menstrual period, whichever is longer, after the last dose of investigational product, agree to have pregnancy tests while in the study and at the end of the study, and agree not to be egg (oocyte) donors while on study and until at least 30 days or 1 menstrual period, whichever is longer, after the last dose of investigational product.
* Sexually active males with female partners who are WOCBP must agree to use two forms of contraception, one of which must be barrier contraception, from screening through 90 days after their last dose of study treatment. All non-sterile male participants must agree not to donate sperm or attempt conception from screening through 90 days following their last dose of study treatment.
* Participants should have ability to understand the purpose and risks of the trial, willingness and ability to comply with the protocol, and provided written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

* Participants with clinically atypical and/or rapidly changing AK lesions in the TF; hyperkeratotic or hypertrophic lesions, recalcitrant disease (defined as failure to respond to cryosurgery on 2 previous occasions) and/or cutaneous horn; history of invasive SCC, Bowen's disease, BCC, or other malignant tumors in the TF; any other dermatological disease that causes difficulty with examination.
* Location of the TF is on any location other than the face or balding scalp, within 5 centimeter (cm) of an incompletely healed wound, within 5 cm of a suspected BCC or other neoplasms, periorbital, lips, or nostrils.
* Participants having a previous treatment with tirbanibulin 10 mg/g ointment.
* Females who are pregnant or nursing or seeking to become pregnant.
* Participants having intention to use any concomitant medication that is not permitted by this protocol or failure to undergo the required washout period for a particular prohibited medication or therapy.
* Participants with anticipated need for inpatient hospitalization or inpatient surgery from Day 1 to Day 113.
* Participants with history of sensitivity and/or allergy to any of the ingredients in the study medication.
* Participants with significant abnormalities on the medical history, physical examination (PE) findings, vital signs, clinical chemistry, or hematology results that in the judgment of the investigator may interfere with the interpretation of the results.
* Participants with skin disease (example; atopic dermatitis, psoriasis, eczema) or condition (example; scarring, open wounds) that, in the opinion of the investigator, might interfere with the study conduct or evaluations, or which exposes the participant to unacceptable risk by study participation.
* Participants with significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the investigator, would expose the participant to unacceptable risk by study participation.
* Participants who have participated in an investigational drug trial during which an investigational study medication was administered within 30 days or 5 half-lives of the investigational product, whichever is longer, before dosing in the current study.
* Participant who is employee or a relative to an employee at the research site or the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline in Lesion Count at Day 57 | Baseline, Day 57
  Percentage change from baseline in the AK lesion count will be assessed.

SECONDARY OUTCOMES:
Proportion of Participants With Partial Clearance (PC) at Day 57 | At Day 57
  PC is defined as proportion of participants achieving more than or equal to (>=) 75 percent (%) clearance of AK lesions in the TF on the face or scalp at Day 57.
Proportion of Participants With Complete Clearance (CC) at Day 57 | At Day 57
  CC is defined as proportion of participants achieving 100 percent clearance of AK lesions in the TF on the face or scalp at Day 57.
Proportion of Participants With Partial Clearance (PC) by Day 113 | Baseline up to Day 113
Proportion of Participants With Complete Clearance (CC) by Day 113 | Baseline up to Day 113
Total Number of Lesions per Participant in the TF at Specific Timepoints | Baseline, Day 8, 15, 29, 57, 64, 71, 85, and 113
Percent Change From Baseline in lesion count in the TF at Specific Timepoints | Baseline, Day 8, 15, 29, 57, 64, 71, 85, and 113
Number of New Lesions per Participant in the TF at Specific Timepoints | At Day 8, 15, 29, 57, 64, 71, 85, and 113
  Number of new lesions that are not present at baseline, occurring per participant in the TF at specific timepoints will be assessed.
Number of Baseline Lesions per Participant Present in the TF at Specific Timepoints | Baseline, Day 8, 15, 29, 57, 64, 71, 85, and 113
  Number of lesions per participant in the TF at specific timepoints will be assessed.
Change From Baseline in Skindex-16 Questionnaire Overall Score and Domain Scores (Symptoms, Emotions, and Functioning) at Day 57 | Baseline, Day 57
  Skindex-16 is used for participants to rate skin conditions that have occurred within the previous week. It is a short 16-item patient-completed assessment that are classified into three domains: symptoms [four items, 1-4], emotions, [seven items, 5-11] and functioning [five items, 12-16]. All items are scored on a seven-point numerical analogue scales (0=never bothered to 6=always bothered). Each item is then transformed to a linear scale from 0 (never bothered) to 100 (always bothered), where higher the score = more severe in impairment. The total score is the average of all 16 items scores ranging from 0 [best Health Related Quality of Life (HRQoL)] to 96 (worst HRQoL), where higher score indicates worst quality of life.
Change from Baseline in Skindex-16 Questionnaire Overall Score and Domain Scores (Symptoms, Emotions, and Functioning) at Day 113 in Participants who Receive 2 Treatment Courses | Baseline, Day 113
  Skindex-16 is used for participants to rate skin conditions that have occurred within the previous week. It is a short 16-item patient-completed assessment that are classified into three domains: symptoms [four items, 1-4], emotions, [seven items, 5-11] and functioning [five items, 12-16]. All items are scored on a seven-point numerical analogue scales (0=never bothered to 6=always bothered). Each item is then transformed to a linear scale from 0 (never bothered) to 100 (always bothered), where higher the score = more severe in impairment. The total score is the average of all 16 items scores ranging from 0 [best Health Related Quality of Life (HRQoL)] to 96 (worst HRQoL), where higher score indicates worst quality of life.
Cosmetic Outcome as Assessed by the Participant at Day 57 | At Day 57
  Cosmetic Outcome is rated on a 4-point scale as excellent (no or mild redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight-to-moderate scarring, atrophy, or induration), and poor (extensive scarring, atrophy, or induration).
Cosmetic Outcome as Assessed by the Investigator at Day 57 | At Day 57
  Cosmetic Outcome is rated on a 4-point scale as excellent (no or mild redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight-to-moderate scarring, atrophy, or induration), and poor (extensive scarring, atrophy, or induration).
Cosmetic Outcome in Participants who Receive 2 Treatment Courses, as Assessed by Participants at Day 113 | At Day 113
  Cosmetic Outcome is rated on a 4-point scale as excellent (no or mild redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight-to-moderate scarring, atrophy, or induration), and poor (extensive scarring, atrophy, or induration).
Cosmetic Outcome in Participants who Receive 2 Treatment Courses, as Assessed by Investigator at Day 113 | At Day 113
  Cosmetic Outcome is rated on a 4-point scale as excellent (no or mild redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight-to-moderate scarring, atrophy, or induration), and poor (extensive scarring, atrophy, or induration).
Treatment Satisfaction Questionnaire for Medications (TSQM) Transformed Total Scores at Day 57 | At Day 57
  The TSQM-14 is a participant-rated scale used to assess subjective satisfaction with medication. The TSQM-14 provided scores on 4 domains: effectiveness (questions 1 to 3) side effects (4 to 8), convenience (9 to 11), and global satisfaction (12 to 14). With the exception of item 4 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied). Scores for each domain were transformed into a final score ranging from 0 to 100, with higher numbers indicating a higher level of satisfaction.
TSQM Transformed Scores in Participants who Receive 2 Treatment Courses at Day 113 | At Day 113
  The TSQM-14 is a participant-rated scale used to assess subjective satisfaction with medication. The TSQM-14 provided scores on 4 domains: effectiveness (questions 1 to 3) side effects (4 to 8), convenience (9 to 11), and global satisfaction (12 to 14). With the exception of item 4 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied). Scores for each domain were transformed into a final score ranging from 0 to 100, with higher numbers indicating a higher level of satisfaction.
Local Tolerability Score at Specific Timepoints for Each Individual Sign | At Day 1, 8, 15, 29, 57, 64, 71, 85, and 113
  Local tolerability score is evaluated by the investigator in terms of presence and absence of erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration signs and its severity in the areas of body where medication is applied. These symptoms are assessed by using a 4-point scale of 0-3, where 0 (absent) and 3 (severe). The higher score indicates severe symptoms.
Maximum Local Tolerability Score in Treatment Course for Each Individual Sign | At Day 1, 8, 15, 29, 57, 64, 71, 85, and 113
  Maximum local tolerability score by treatment course for each individual sign (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) will be assessed. Local tolerability score for each signs are assessed by using a 4 - point scale of 0 - 3, where 0 = none and 3 = severe. The higher score indicates severe symptoms.
Time to Maximum Local Tolerability Score Observed in Treatment Course for Each Individual Sign | At Day 1, 8, 15, 29, 57, 64, 71, 85, and 113
  Time to maximum local tolerability score for erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration will be assessed. Maximum local tolerability score by treatment course for each individual sign (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) will be assessed. Local tolerability score for each signs are assessed by using a 4 - point scale of 0 - 3, where 0 = none and 3 = severe. The higher score indicates severe symptoms.
Local Tolerability Signs Composite Score at Specific Timepoints | At Day 1, 8, 15, 29, 57, 64, 71, 85, and 113
  Local tolerability signs composite score (0-18) at Specific Timepoints, defined as the sum of the scores graded from 0 (none) to 3 (severe) on all six individual tolerability sign categories (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) will be assessed. The higher score indicates severe symptoms.
Maximum Local tolerability Signs Composite Score in Treatment Course | At Day 1, 8, 15, 29, 57, 64, 71, 85, and 113
  Maximum local tolerability signs composite score (0-18) in treatment course, defined as the sum of the scores graded from 0 (none) to 3 (severe) on all six individual tolerability sign categories (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) will be assessed. The higher score indicates severe symptoms.
Time to Maximum Local Tolerability Signs Composite Score Observed in Treatment Course | At Day 1, 8, 15, 29, 57, 64, 71, 85, and 113
  Time to maximum local tolerability signs composite score is observed in treatment course for each individual sign (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) will be assessed. Maximum local tolerability signs composite score (0-18) in treatment course, defined as the sum of the scores graded from 0 (none) to 3 (severe) on all six individual tolerability sign categories (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) will be assessed. The higher score indicates severe symptoms.
Number of Participants Showing Changes in Pigmentation and Scarring in the TF at Specific Timepoints | At Day 1, 8, 15, 29, 57, 64, 71, 85, and 113
  Absence or presence of pigmentation (that is, hypopigmentation and hyperpigmentation) and scarring in the TF will be assessed.
Number of Participants With Adverse Event (AE), Serious Adverse Events (SAEs) and Adverse Events of Special Interests (AESIs) | From Screening up to Day 113
  An AE is defined as any untoward medical occurrence in a clinical trial participant, regardless of the administration of the IMP and its causal relationship to it. unfavorable and unintended medical occurrence during the participant's participation in the trial, including deterioration of a pre-existing medical condition, an abnormal value in a laboratory assessment, or an abnormal finding in the physical examination. An SAE is any untoward medical occurrence that at any dose resulted in death; is life threatening; required persistent/significant disability/incapacity; resulted in initial or prolonged in participant hospitalization; is congenital anomaly/birth defect or otherwise considered medically important. AESIs included skin cancers [including basal cell carcinoma (BCC), squamous cell carcinoma (SCC), and melanoma] appearing within or outside the TF during the study.
Number of Participants With Clinically Significant Laboratory Abnormalities | From Screening up to Day 113
  Number of participants with clinically significant laboratory abnormalities (included hematology, blood chemistry and urinalysis) will be assessed. Clinically Significant Abnormal values will be determined by the investigator.
Number of Participants With Vital Signs Abnormalities | From Screening up to Day 113
  Number of participants with vital signs (including measurement of systolic and diastolic blood pressure, heart rate, respiratory rate, and tympanic temperature) will be assessed. Abnormal values will be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (35):
- Germany (8):
  - Site 17, Augsburg
  - Site 1, Bad Bentheim
  - Site 3, Bochum
  - Site 18, Dresden
  - Site 2, Hamburg
  - Site 5, Hamburg
  - Site 4, Mahlow
  - Site 6, Wuppertal
- Italy (10):
  - Site 24, Bari
  - Site 25, Bologna
  - Site 19, Brescia
  - Site 26, Cagliari
  - Site 23, Florence
  - Site 22, Pisa
  - Site 27, Reggio Emilia
  - Site 20, Roma
  - Site 21, Roma
  - Site 7, Roma
- Netherlands (2):
  - Site 29, Heemstede
  - Site 28, Maastricht
- Poland (6):
  - Site 31, Krakow
  - Site 30, Ossy
  - Site 10, Warsaw
  - Site 11, Warsaw
  - Site 9, Warsaw
  - Site 8, Wroclaw
- Spain (9):
  - Site 12, Barcelona
  - Site 14, Barcelona
  - Site 34, Barcelona
  - Site 33, Granada
  - Site 13, Madrid
  - Site 32, Salamanca
  - Site 15, Valencia
  - Site 35, Valencia
  - Site 16, Zaragoza

IPD SHARING:
Plan to Share IPD: No